CLINICAL TRIAL: NCT07097285
Title: The Effect of Sensory Awareness Training Given to Women of Reproductive Age on Dysmenorrhea and Kinesiophobia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Doç. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SBÜ-AYDINKARTAL-015
Record Dates: First submitted 2024-12-08; First posted 2025-07-31 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Dysmenorrhea; Kinesiophobia
Keywords: Sensory Awareness; Dysmenorrhea; Kinesiophobia; Reproductive; Women
MeSH Terms: conditions — Dysmenorrhea; Kinesiophobia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care (n:40) (No Intervention): No intervention will be made to the control group.
- sensory awareness training (n:40) (Experimental): Sensory awareness training was given to women in the intervention group of the study for 4 weeks. will be given. Each training is 60 minutes long will be planned. 4 weeks from pre-training and first training "Tampa Kinesiophobia Scale (TKÖ)" "Dysmenorrhea Affectedness Scale" and "Very Dimensional Body Awareness Assessment-II Scale" will be applied. be once a week Each training period is limited to 60 minutes. Research forms were given to participants face to face. will be implemented.
  Interventions: Behavioral: sensory awareness training

INTERVENTIONS:
Behavioral: sensory awareness training — Presentations to inform during training will be done, then Graded Sensory Discrimination, Graded Motor Imagery (DMI) and a home exercise program, as well as a body awareness training program. protocol will be applied. Graded Sensory Discrimination protocol, localization training It includes level 1, localization training level 2 and graphesthesia training. Graded Engine Visualization (DMI) protocol includes right/left discrimination training and visual imagery training.
  Arms: sensory awareness training (n:40)

SUMMARY:
This research investigates the use of web-based sensory awareness training given to women of reproductive age. It was planned to examine the effect of dysmenorrhea level and kinzeophobia status.H0a = Body weight of women of reproductive age who received and did not receive sensory awareness training. There is no difference between awareness levels.

H1a = Body size of women of reproductive age who receive and do not receive sensory awareness training. There is a difference between awareness levels.

H0b = Dysmenorrhea of women of reproductive age who received or did not receive sensory awareness training. There is no difference between the levels.

H1b = Dysmenorrhea among women of reproductive age who received and did not receive sensory awareness training. There is a difference between the levels.

H0c = Kinesiophobia in women of childbearing age who received or did not receive sensory awareness training. There is no difference between the situations.

H1c = Kinesiophobia in women of reproductive age who receive and do not receive sensory awareness training. There is a difference between situations Sensory awareness training was given to women in the intervention group of the study for 4 weeks. will be given. Training contents, Sensory System Training Presentation, Proprioception and Kinesthesia Sensory Training Presentation, Interoception Sense Training Presentation will be given, then Graded Sensory Discrimination, Graded Motor Imagery (DMI), interoception awareness training, body training with training consisting of interoceptive awareness exercises and home exercise programs. A protocol for awareness training will be implemented.

DETAILED DESCRIPTION:
Sensory awareness training was given to women in the intervention group of the study for 4 weeks will be given. Training contents, Sensory System Training Presentation, Proprioception and Kinesthesia Sensory Training Presentation, Interoception Sense Training Presentation will be given, then Graded Sensory Discrimination, Graded Motor Imagery (DMI), interoception awareness training, body training with training consisting of interoceptive awareness exercises and home exercise programs.

A protocol for awareness training will be implemented. Each training is 60 minutes long will be planned. Women who volunteered to participate in the study and were assigned to the intervention group An informational meeting will be held before the training. 4 weeks from pre-training and first training "Tampa Kinesiophobia Scale (TKÖ)" "Dysmenorrhea Affectedness Scale" and "Very Dimensional Body Awareness Assessment-II Scale" will be applied. be once a week Each training period is limited to 60 minutes. Research forms were given to participants face to face. will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in research
* Having a complaint of dysmonea
* Being of childbearing age
* Being over 19 years old
* Having internet access
* Having a smart mobile phone

Exclusion Criteria:

* Be pregnant
* Having any disease that affects the menstrual period
* Using oral contraceptives
* Using intrauterine device

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | Baseline
  In this form created by researchers based on the literature, There are questions about the participants' age, the high school they graduated from, dysmenorrhea and kinesiophobia is taking.
Tampa Kinesiophobia Scale | day 1
  Tampa Kinesiophobia Scale (TCS) Miller, Kori and Todd It is a scale developed by in 1991. Fear of movement and re-injury, and It was developed to evaluate avoidance behavior due to fear. It was adapted to Turkish by Yılmaz et al. in 2011 and tested for validity and reliability. study has been done. The scale consists of 17 questions. On the scale, "1" means "strongly disagree" and "2" means "strongly disagree." from "1" to "4", where "I disagree", "3" I agree, "4" I completely agree. Varying Likert scoring is used. An individual can get a total score between 17-68, A high score indicates that the individual has high kinesiophobia.
Dysmenorrhea Affect Scale | day 1
  Validity and reliability study by Gün (2014) The Dysmenorrhea Exposure Scale (DES) was used to measure women's periods of menstrual pain. It is designed to identify problems and coping methods. A total of items 39 and 11 It consists of sub-dimensions. The Cronbach's Alpha coefficient of the scale is 0.90. Participants each rated the item on a 5-point scale ranging from 'I totally disagree (1)' to 'I totally agree (5)'. It evaluates on a Likert type scale. As the score obtained from the scale increases, people's The level of being affected by dysmenorrhea also increases. The lowest score that can be obtained from the scale is , The highest score is 195.
Multidimensional Body Awareness Assessment-II Scale | day 1
  Body Awareness has multiple developed by Mehling, Acree, Stewart, Silas and Jones to measure the dimensions of The Turkish adaptation of the scale was made by Mungurlar and Kahya. Scale, It is a self-report scale consisting of one item and eight factors. These factors; "Noticing", "Attention "Not Distracting", "Not Worrying", "Regulating Attention", "Emotional Awareness", "Self-Regulation", "Listening to the Body" and "Trusting". Evaluation of the scale is 1-5 points and is made by averaging the scoring factors separately. of scale Validity reliability Cronbach's alpha coefficient was determined as 0.88. As the score obtained from the scale increases, it means that people have more positive body awareness.

SECONDARY OUTCOMES:
Tampa Kinesiophobia Scale | up to 4 weeks
  Tampa Kinesiophobia Scale (TCS) Miller, Kori and Todd It is a scale developed by in 1991. Fear of movement and re-injury, and It was developed to evaluate avoidance behavior due to fear. It was adapted to Turkish by Yılmaz et al. in 2011 and tested for validity and reliability. study has been done. The scale consists of 17 questions. On the scale, "1" means "strongly disagree" and "2" means "strongly disagree." from "1" to "4", where "I disagree", "3" I agree, "4" I completely agree. Varying Likert scoring is used. An individual can get a total score between 17-68, A high score indicates that the individual has high kinesiophobia.
Dysmenorrhea Affect Scale | up to 4 weeks
  Validity and reliability study by Gün (2014) The Dysmenorrhea Exposure Scale (DES) was used to measure women's periods of menstrual pain. It is designed to identify problems and coping methods. A total of items 39 and 11 It consists of sub-dimensions. The Cronbach's Alpha coefficient of the scale is 0.90. Participants each rated the item on a 5-point scale ranging from 'I totally disagree (1)' to 'I totally agree (5)'. It evaluates on a Likert type scale. As the score obtained from the scale increases, people's The level of being affected by dysmenorrhea also increases. The lowest score that can be obtained from the scale is , The highest score is 195.
Multidimensional Body Awareness Assessment-II Scale | up to 4 weeks
  Body Awareness has multiple developed by Mehling, Acree, Stewart, Silas and Jones to measure the dimensions of The Turkish adaptation of the scale was made by Mungurlar and Kahya. Scale, It is a self-report scale consisting of one item and eight factors. These factors; "Noticing", "Attention "Not Distracting", "Not Worrying", "Regulating Attention", "Emotional Awareness", "Self-Regulation", "Listening to the Body" and "Trusting". Evaluation of the scale is 1-5 points and is made by averaging the scoring factors separately. of scale Validity reliability Cronbach's alpha coefficient was determined as 0.88. As the score obtained from the scale increases, it means that people have more positive body awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi, Istanbul, Turkey (Türkiye)